CLINICAL TRIAL: NCT04213963
Title: Prospective Cross-sectional Study on Prevalence of Primary Aldosteronism in Resistant Hypertension and Association With Cardiometabolic Complications
Brief Title: Prospective Study on Primary Aldosteronism in Resistant Hypertension
Acronym: PrePARe
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Mauro Maccario, Medical Doctor, Professor, University of Turin, Italy
Other Study IDs: The PrePARe Study
Record Dates: First submitted 2019-12-19; First posted 2019-12-30 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Resistant Hypertension; Primary Aldosteronism; Refractory Hypertension; Hypertensive End-Organ Damage; Atrial Fibrillation; Aortic Ectasia
Keywords: Resistant Hypertension; Primary Aldosteronism; Renin-Angiotensin System; Blood Pressure; Cardiometabolic Risk; Early Atherosclerotic Damage; Oxidative Stress
MeSH Terms: conditions — Hyperaldosteronism; Hypertension; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood (5), plasma (1), serum (11) and salivary samples (2) with 24-hour urine collection (1).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prevalence of primary aldosteronism (PA) in resistant hypertension is not clear. In addition, emerging evidence supports the role of elevated serum aldosterone in promoting cardiovascular disease, independently from high blood pressure (BP) levels, but current data on this issue are heterogeneous.

DETAILED DESCRIPTION:
PA is the most frequent form of secondary hypertension, with a prevalence that increases with the severity of hypertension. The wide variation of the reported PA prevalence is due to different study design and population. Very few data derive from well designed prospective study. Additional problems in the interpretation of study results are the different diagnostic cut-off used in various centers and the low diffusion of the adrenal vein sampling, that has a central role in the PA diagnosis.

Resistant hypertension (RH) is a condition of insufficient BP control, despite appropriate lifestyle measures and treatment with at least 3 drugs at full dose, including a diuretic, in patients whose adherence to therapy has been confirmed. The primary aim of our study is define prospectively the prevalence of PA in RH.

Moreover, emerging evidence supports the crucial role of elevated serum aldosterone in promoting cardiovascular disease, independently from high BP levels. Aldosterone improves oxidative stress, inflammation, impairs insulin metabolic signaling, reduced endothelial-mediated vasorelaxation and is associated to cardiovascular and renal abnormalities. However, current data on the contribution of PA on cardiometabolic complications have heterogeneous results.

The secondary outcome of our study is to investigate prospectively the association of PA with cardiometabolic complications in a cohort of patients with RH.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 and under 80 years old;
* diagnosis of resistant hypertension defined as: uncontrolled blood pressure at ambulatory blood pressure measurement (ABPM), despite the use of at least 3 antihypertensive drugs at full dose, including a diuretic.

Exclusion Criteria:

* age under 18 or over 80 years old;
* pseudo-resistant hypertension (poor medication adherence, high salt intake);
* previous cardiovascular disease;
* insulin treated diabetes mellitus;
* other than primary aldosteronism cause of secondary hypertension (obstructive sleep apnea, renal artery stenosis, pheochromocytoma/paraganglioma, primary hyperparathyroidism, autonomous cortisol secretion or over hypercortisolism);
* liver cirrhosis;
* chronic heart failure;
* known malignant neoplasm;
* chronic disease with major organ involvement;
* excessive alcohol ingestion;
* current steroids assumption;
* use of sympathomimetic drugs;
* use of contraceptives.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At least 100 consecutive patients with age over 18 and under 80 years old and resistant hypertension (defined as uncontrolled blood pressure despite the use of at least 3 antihypertensive drugs at full dose, including a diuretic) referred to the center for diagnosis and treatment of Hypertension (Division of Endocrinology, Diabetology and Metabolism, University of Turin) between March 2011 and July 2020.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-09-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of diagnosis (prevalence) of primary aldosteronism in prospective cohort of patients with resistant hypertension. | Baseline.
  Basal Aldosterone (pg/mL) at baseline.
Number of diagnosis (prevalence) of primary aldosteronism in prospective cohort of patients with resistant hypertension. | Baseline.
  Basal Plasma Renin Activity (PRA, ng/mL/h) at baseline.
Number of diagnosis (prevalence) of primary aldosteronism in prospective cohort of patients with resistant hypertension. | Baseline.
  Aldosterone (pg/mL) post saline infusion test, performed at baseline.

SECONDARY OUTCOMES:
Left ventricular hypertrophy in primary aldosteronism and essential resistant hypertension | Baseline.
  Left ventricular mass evaluation with Echocardiogram at baseline.
Microalbuminuria in primary aldosteronism and essential resistant hypertension. | Baseline.
  Albuminuria/Creatininuria ratio (mg/mmoL) at baseline.
Intima media thickness > 0.9 mm rate in primary aldosteronism versus essential resistant hypertension. | Baseline
  Intima media thickness values (mm) evaluation with carotid Doppler ultrasound at baseline.
Chronic kidney disease in primary aldosteronism versus essential resistant hypertension. | Baseline.
  Serum creatinine (mg/dL) at baseline.
Aortic ectasia in primary aldosteronism versus essential resistant hypertension. | Baseline.
  Aortic size (mm) determined with echocardiogram at baseline.
Atrial fibrillation in primary aldosteronism versus essential resistant hypertension. | Baseline.
  Electrocardiogram (ECG) at baseline.
Insulin resistance in primary aldosteronism versus essential resistant hypertension. | Baseline
  Oral glucose tolerance test (OGTT) for determination of glucose (mg/dL) at time 0', 30', 60', 90' and 120' at baseline.
Insulin resistance in primary aldosteronism versus essential resistant hypertension. | Baseline.
  Oral glucose tolerance test (OGTT) for determination of insulin (mg/dL) at time 0', 30', 60', 90' and 120' at baseline.
Diabetes mellitus rate in primary aldosteronism versus essential resistant hypertension. | Baseline.
  Oral glucose tolerance test (OGTT) for determination of glucose (mg/dL) at time 0' and 120' at baseline.
Diabetes mellitus rate in primary aldosteronism versus essential resistant hypertension. | Baseline.
  HbA1c (mmol/mol) at baseline.
Sodium levels in primary aldosteronism versus essential resistant hypertension. | Baseline.
  Serum Sodium (mmol/L) at baseline.
Potassium levels in primary aldosteronism versus essential resistant hypertension. | Baseline.
  Serum Potassium (mmol/L) at baseline.
Oxidative stress in primary aldosteronism versus essential resistant hypertension. | Baseline.
  Blood determination of 8-isoprostane (UI/L) at baseline.
Oxidative stress in primary aldosteronism versus essential resistant hypertension. | Baseline.
  Blood determination of total antioxidant capacity (UI/L) at baseline.
Dyslipidemia in primary aldosteronism versus essential resistant hypertension. | Baseline.
  Serum triglycerides (mg/dL) at baseline.
Dyslipidemia in primary aldosteronism versus essential resistant hypertension. | Baseline.
  Serum total-Cholesterol (mg/dL) at baseline.
Dyslipidemia in primary aldosteronism versus essential resistant hypertension. | Baseline.
  Serum HDL-Cholesterol (mg/dL) at baseline.
Dyslipidemia in primary aldosteronism versus essential resistant hypertension. | Baseline.
  Serum LDL-Cholesterol (mg/dL) at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Mauro M Maccario, MD, Principal Investigator — Endocrinology, Diabetology and Metabolism; University of Turin; Ezio E Ghigo, MD, Study Chair — Endocrinology, Diabetology and Metabolism; University of Turin
Locations (1):
- Division of Endocrinology, Diabetology and Metabolism; University of Turin, Turin, Piedmont, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Funder JW, Carey RM, Mantero F, Murad MH, Reincke M, Shibata H, Stowasser M, Young WF Jr. The Management of Primary Aldosteronism: Case Detection, Diagnosis, and Treatment: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2016 May;101(5):1889-916. doi: 10.1210/jc.2015-4061. Epub 2016 Mar 2. PMID 26934393
- [Result] Monticone S, Burrello J, Tizzani D, Bertello C, Viola A, Buffolo F, Gabetti L, Mengozzi G, Williams TA, Rabbia F, Veglio F, Mulatero P. Prevalence and Clinical Manifestations of Primary Aldosteronism Encountered in Primary Care Practice. J Am Coll Cardiol. 2017 Apr 11;69(14):1811-1820. doi: 10.1016/j.jacc.2017.01.052. PMID 28385310
- [Result] Rossi GP, Bernini G, Caliumi C, Desideri G, Fabris B, Ferri C, Ganzaroli C, Giacchetti G, Letizia C, Maccario M, Mallamaci F, Mannelli M, Mattarello MJ, Moretti A, Palumbo G, Parenti G, Porteri E, Semplicini A, Rizzoni D, Rossi E, Boscaro M, Pessina AC, Mantero F; PAPY Study Investigators. A prospective study of the prevalence of primary aldosteronism in 1,125 hypertensive patients. J Am Coll Cardiol. 2006 Dec 5;48(11):2293-300. doi: 10.1016/j.jacc.2006.07.059. Epub 2006 Nov 13. PMID 17161262
- [Result] Mulatero P, Stowasser M, Loh KC, Fardella CE, Gordon RD, Mosso L, Gomez-Sanchez CE, Veglio F, Young WF Jr. Increased diagnosis of primary aldosteronism, including surgically correctable forms, in centers from five continents. J Clin Endocrinol Metab. 2004 Mar;89(3):1045-50. doi: 10.1210/jc.2003-031337. PMID 15001583
- [Result] Calhoun DA, Nishizaka MK, Zaman MA, Thakkar RB, Weissmann P. Hyperaldosteronism among black and white subjects with resistant hypertension. Hypertension. 2002 Dec;40(6):892-6. doi: 10.1161/01.hyp.0000040261.30455.b6. PMID 12468575
- [Result] Strauch B, Zelinka T, Hampf M, Bernhardt R, Widimsky J Jr. Prevalence of primary hyperaldosteronism in moderate to severe hypertension in the Central Europe region. J Hum Hypertens. 2003 May;17(5):349-52. doi: 10.1038/sj.jhh.1001554. PMID 12756408
- [Result] Eide IK, Torjesen PA, Drolsum A, Babovic A, Lilledahl NP. Low-renin status in therapy-resistant hypertension: a clue to efficient treatment. J Hypertens. 2004 Nov;22(11):2217-26. doi: 10.1097/00004872-200411000-00026. PMID 15480108
- [Result] Chandran P. Resistant or difficult-to-control hypertension. N Engl J Med. 2006 Nov 2;355(18):1934; author reply 1934. doi: 10.1056/NEJMc062276. No abstract available. PMID 17079772
- [Result] Schmidt BM, Schmieder RE. Aldosterone-induced cardiac damage: focus on blood pressure independent effects. Am J Hypertens. 2003 Jan;16(1):80-6. doi: 10.1016/s0895-7061(02)03199-0. PMID 12517689
- [Result] Fallo F, Veglio F, Bertello C, Sonino N, Della Mea P, Ermani M, Rabbia F, Federspil G, Mulatero P. Prevalence and characteristics of the metabolic syndrome in primary aldosteronism. J Clin Endocrinol Metab. 2006 Feb;91(2):454-9. doi: 10.1210/jc.2005-1733. Epub 2005 Nov 15. PMID 16291704
- [Result] Rossi GP, Sechi LA, Giacchetti G, Ronconi V, Strazzullo P, Funder JW. Primary aldosteronism: cardiovascular, renal and metabolic implications. Trends Endocrinol Metab. 2008 Apr;19(3):88-90. doi: 10.1016/j.tem.2008.01.006. Epub 2008 Mar 7. PMID 18314347
- [Result] Whaley-Connell A, Johnson MS, Sowers JR. Aldosterone: role in the cardiometabolic syndrome and resistant hypertension. Prog Cardiovasc Dis. 2010 Mar-Apr;52(5):401-9. doi: 10.1016/j.pcad.2009.12.004. PMID 20226958
- [Result] Fiebeler A, Luft FC. The mineralocorticoid receptor and oxidative stress. Heart Fail Rev. 2005 Jan;10(1):47-52. doi: 10.1007/s10741-005-2348-y. PMID 15947891
- [Result] Vogt B, Burnier M. Aldosterone and cardiovascular risk. Curr Hypertens Rep. 2009 Dec;11(6):450-5. doi: 10.1007/s11906-009-0076-8. PMID 19895757
- [Result] Morrow JD. Quantification of isoprostanes as indices of oxidant stress and the risk of atherosclerosis in humans. Arterioscler Thromb Vasc Biol. 2005 Feb;25(2):279-86. doi: 10.1161/01.ATV.0000152605.64964.c0. Epub 2004 Dec 9. PMID 15591226
- [Result] Prior RL, Cao G. In vivo total antioxidant capacity: comparison of different analytical methods. Free Radic Biol Med. 1999 Dec;27(11-12):1173-81. doi: 10.1016/s0891-5849(99)00203-8. PMID 10641708
- [Result] Vassalle C, Pratali L, Boni C, Mercuri A, Ndreu R. An oxidative stress score as a combined measure of the pro-oxidant and anti-oxidant counterparts in patients with coronary artery disease. Clin Biochem. 2008 Oct;41(14-15):1162-7. doi: 10.1016/j.clinbiochem.2008.07.005. Epub 2008 Jul 26. PMID 18692492
- [Result] Fallo F, Della Mea P, Sonino N, Bertello C, Ermani M, Vettor R, Veglio F, Mulatero P. Adiponectin and insulin sensitivity in primary aldosteronism. Am J Hypertens. 2007 Aug;20(8):855-61. doi: 10.1016/j.amjhyper.2007.03.012. PMID 17679033
- [Result] Iacobellis G, Petramala L, Cotesta D, Pergolini M, Zinnamosca L, Cianci R, De Toma G, Sciomer S, Letizia C. Adipokines and cardiometabolic profile in primary hyperaldosteronism. J Clin Endocrinol Metab. 2010 May;95(5):2391-8. doi: 10.1210/jc.2009-2204. Epub 2010 Mar 1. PMID 20194710
- [Result] Giacchetti G, Sechi LA, Rilli S, Carey RM. The renin-angiotensin-aldosterone system, glucose metabolism and diabetes. Trends Endocrinol Metab. 2005 Apr;16(3):120-6. doi: 10.1016/j.tem.2005.02.003. PMID 15808810
- [Result] Lucatello B, Benso A, Tabaro I, Capello E, Caprino MP, Marafetti L, Rossato D, Oleandri SE, Ghigo E, Maccario M. Long-term re-evaluation of primary aldosteronism after medical treatment reveals high proportion of normal mineralocorticoid secretion. Eur J Endocrinol. 2013 Mar 15;168(4):525-32. doi: 10.1530/EJE-12-0912. Print 2013 Apr. PMID 23321497
- [Result] Rossi GP, Maiolino G, Flego A, Belfiore A, Bernini G, Fabris B, Ferri C, Giacchetti G, Letizia C, Maccario M, Mallamaci F, Muiesan ML, Mannelli M, Negro A, Palumbo G, Parenti G, Rossi E, Mantero F; PAPY Study Investigators. Adrenalectomy Lowers Incident Atrial Fibrillation in Primary Aldosteronism Patients at Long Term. Hypertension. 2018 Apr;71(4):585-591. doi: 10.1161/HYPERTENSIONAHA.117.10596. Epub 2018 Feb 26. PMID 29483224
- [Result] Douma S, Petidis K, Doumas M, Papaefthimiou P, Triantafyllou A, Kartali N, Papadopoulos N, Vogiatzis K, Zamboulis C. Prevalence of primary hyperaldosteronism in resistant hypertension: a retrospective observational study. Lancet. 2008 Jun 7;371(9628):1921-6. doi: 10.1016/S0140-6736(08)60834-X. PMID 18539224
- [Result] Marzano L, Colussi G, Sechi LA, Catena C. Adrenalectomy is comparable with medical treatment for reduction of left ventricular mass in primary aldosteronism: meta-analysis of long-term studies. Am J Hypertens. 2015 Mar;28(3):312-8. doi: 10.1093/ajh/hpu154. Epub 2014 Oct 21. PMID 25336498